CLINICAL TRIAL: NCT05854953
Title: A Randomised Crossover Clinical Trial to Compare the Effects of Different Storage Conditions on Removable Retainers
Brief Title: The Effects of Different Storage Conditions on Removable Retainers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Wan Nurazreena Wan Hassan, Associate Professor, Department of Paediatric Dentistry & Orthodontics, Faculty of Dentistry, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: S2042680
Record Dates: First submitted 2023-04-17; First posted 2023-05-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Orthodontic Appliance Complication
Keywords: removable retainers; wet storage condition; dry storage condition

STUDY DESIGN:
Intervention Model Description: Baseline characteristics - newly constructed Hawley and vacuum-formed retainers will be tested for microbial analysis, phyiscal and mechanical properties as comparisons with other groups
  Group 1 - Participants with Hawley retainers will begin storing their retainers in dry condition, 3 months later, they will change the storage to wet condition.
  Group 2 - Participants with Hawley retainers will begin storing their retainers in wet condition, 3 months later, they will change the storage to dry condition.
  Group 3 - Participants with vacuum-formed retainers will begin storing their retainers in dry condition, 3 months later, they will change the storage to wet condition.
  Group 4 - Participants with vacuum-formed retainers will begin storing their retainers in wet condition, 3 months later, they will change the storage to dry condition.
Who Masked: Investigator
Masking Description: Investigator will be masked with the randomization sequance & allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Hawley retainers in dry storage condition (Experimental): Acrylic retainers to be stored in a dry retainer box the entire time when not in use.
  Interventions: Device: Hawley retainers in dry storage condition
- Hawley retainers in wet storage condition (Experimental): Acrylic retainers to be stored in a glass of clean tap water the entire time when not in use.
  Interventions: Device: Hawley retainers in wet storage condition
- Vacuum-formed retainers in dry storage condition (Experimental): Thermoplastic retainers to be stored in a dry retainer box the entire time when not in use.
  Interventions: Device: VFRs in dry storage condition
- Vacuum-formed retainers in wet storage condition (Experimental): Thermoplastic retainers to be stored in a glass of clean tap water the entire time when not in use.
  Interventions: Device: VFRs in wet storage condition
- Baseline characteristics (Active Comparator): Newly constructed Hawley retainers and VFRs will be labeled as baseline samples.
  Interventions: Device: Baseline characteristics

INTERVENTIONS:
Device: Hawley retainers in dry storage condition — Three months later, an exchange of storage methods from dry to wet conditions will take place.
  Other Names: Acrylic retainers
  Arms: Hawley retainers in dry storage condition
Device: Hawley retainers in wet storage condition — Three months later, an exchange of storage methods from wet to dry conditions will take place.
  Other Names: Acrylic retainers
  Arms: Hawley retainers in wet storage condition
Device: VFRs in dry storage condition — Three months later, an exchange of storage methods from dry to wet conditions will take place.
  Other Names: Thermoplastic clear retainers
  Arms: Vacuum-formed retainers in dry storage condition
Device: VFRs in wet storage condition — Three months later, an exchange of storage methods from wet to dry conditions will take place.
  Other Names: Thermoplastic clear retainers
  Arms: Vacuum-formed retainers in wet storage condition
Device: Baseline characteristics — Hawley retainers and VFRs that are newly constructed will be used as baseline samples. The samples will be taken for microbial, physical and mechanical tests.
  Arms: Baseline characteristics

SUMMARY:
Orthodontic removable retainers are appliances that hold the position of the upper and lower teeth after fixed braces treatment and they can be removed from a patient's mouth. Basically, there are 2 types of removable retainers; Hawley retainer and vacuum-formed retainer.

Hawley retainer is made of an acrylic resin plate that covers the palate for the upper jaw and the back of the arch facing the tongue for the lower jaw. It has thin stainless-steel wires incorporated to fit the first molars and the six front teeth as retention.

Vacuum-formed retainer (VFR) is a clear or transparent plastic retainer. It covers the teeth completely and a small part of the gum.

The investigators' interest is to determine whether the storage conditions will affect the amount of bacteria, appearance and strength of removable retainers. Primarily, the amount of bacteria that sticks to the retainers may cause overall dental and oral health effects such as mouth odour, dental caries and gum problems. The investigators would also like to assess the oral health-related quality of life (OHRQoL) of participants after storing retainers in different storage conditions by answering a questionnaire.

DETAILED DESCRIPTION:
RATIONALE OF THE STUDY

A non-bias clinical study is required to facilitate the best recommendation to care for the orthodontic retainers. This may prevent the risk of further harms to the oral condition and increase the longevity of the retainers. In turn, this would improve the OHRQoL of orthodontic patients and potentially save the cost of retainer replacements. Therefore, the findings may help to provide evidence-based guidelines for the storage method of removable retainers.

Primary Objective

1. To compare the microbial colony counts of removable retainers in wet and dry storage conditions.

   Secondary Objectives
2. To compare the surface roughness of removable retainer materials in wet and dry storage conditions.
3. To compare the colour stability of removable retainer materials in wet and dry storage conditions.
4. To compare the compressive strength of removable retainer materials in wet and dry storage conditions.
5. To evaluate OHRQoL of participants storing their removable retainers in dry and wet conditions.

SAMPLE SIZE CALCULATION

Sample size calculation was done using G* Power 3.1. The total sample size is 18, for an alpha error equivalent to 0.05, a study power equivalent to 80%, a two-sided test type, and an effect size of 1.316 (Farhadian et al., 2016). Considering a potential dropout of 30%, therefore 24 participants will be recruited.

METHODOLOGY

Participants who fit the inclusion and exclusion criteria will be invited to enrol at the Orthodontic Postgraduate Clinic, Faculty of Dentistry, Universiti Malaya. Once the participants consent to take part in this study, an explanation will be given in detail of the procedure of the research with the aid of the flowchart diagram. The participants will also be given a participant information sheet. An appointment for the removal of fixed braces will be scheduled.

All participants will be required to draw lots from the sealed envelope which has been randomised by the consultant orthodontist to know their first retainer storage condition. The investigator will have to check the group allocation with the consultant orthodontist.

On the first appointment day, the removal of braces will be done according to the standard protocol. Then, four sets of impressions will be taken to construct the models and retainers. The participants will be issued with their regular upper and lower retainers, a new toothbrush and a retainer box. The participants will be instructed to store their retainers in a dry retainer box or in a glass of clean water the entire time when not in use. Other home care instructions include: 1) wear the retainers part-time (8-12 hours daily), 2) clean the retainers with a soft-bristled toothbrush and rinse thoroughly, and 3) no additional cleaning solutions and tablets are allowed. The participants will need to answer a self-administered questionnaire 1 week later to assess their personal judgment on the removable retainers.

The participants will be called 3 months later for review (T1). During this visit, the standard retainers will be taken by the investigator for analysis. The interventional retainers will be issued to the participants with an instruction to exchange the storage method from dry to wet conditions and from wet to dry conditions. The same home care instructions will be advised. The participants will receive a new toothbrush to clean their appliance and a new retainer box to keep their retainers. The participants will need to answer a questionnaire sheet again.

The participants will be called 6 months later for review (T2). The first interventional retainers will be taken by the investigator for the final analysis. The second interventional retainers will be issued to the participants and they will be instructed to continue caring for their retainers. All participants will be required to answer a questionnaire sheet for the final time.

Three different sets of the newly constructed Hawley and vacuum-formed retainers will be tested for microbial analysis, physical and mechanical properties as baseline characteristics for comparisons.

STATISTICAL ANALYSIS

Results obtained will be computed using SPSS Statistics for Windows, Version 26.0. Statistical significance will be set at p < 0.05.

The manipulating variables are the types of storage conditions, which are dry and wet with α = 5% = 0.05 and confidence interval (CI) of 95%. Test of normality will be done using the Shapiro-Wilk test for each of the dependent variables (outcomes).

i. Mann-Whitney U-Test will be applied to compare the dependent variables of the two groups (Hawley retainers and VFRs) at baseline, T1 and T2.

ii. Wilcoxon Signed Rank test will be used to compare the storage conditions of the two groups (Hawley retainers and VFRs) at baseline, T1 and T2.

iii. Kruskal Wallis will be carried out to investigate the interaction between the two samples and the storage conditions.

iv. If the data is normally distributed, then the equivalent parametric analyses (paired t-test and independent t-test) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Fixed appliance treatment on both the upper and lower arches
* Ready for debond
* Planned for either Hawley retainers or VFRs for retention
* Fit and healthy patients without systemic disease
* Non-smoking patients

Exclusion Criteria:

* Sectional fixed appliance treatment or fixed appliance treatment on single arch only
* Planned for double retention with bonded retainers
* Systemic disease that may affect salivary flow
* Smoking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Microbial colony counts of removable retainers in wet and dry storage conditions | 6 months
  Removable retainers will be sonicated and vortexed to dislodge bacteria. Serial dilution will be done and bacterial suspension will be pipetted on a BHI agar petri dish. Total bacterial count in CFU/ml will be counted at baseline, T1 and T2.

SECONDARY OUTCOMES:
Surface roughness of removable retainers in wet and dry storage conditions | 6 months
  Surface roughness will be measured with a surface roughness profilometer (Mitutoyo, Japan). A stylus will make a contact on a surface of the removable retainer and give a measurement in Ra (average surface roughness) parameter. Reading will be taken at baseline, T1 and T2.
Colour stability of removable retainers in wet and dry storage conditions | 6 months
  The colour changes of the removable retainers will be measured with a colour spectrophotometer (Konica Minolta, Japan) at baseline, T1 and T2.
Compressive strength of removable retainers in wet and dry storage conditions | 6 months
  Compressive strength will be done using a universal testing machine (AG-X Series, Shimadzu, Japan). 5 kN compressive load with a loading rate of 1.0 mm/min will be applied at baseline, T1 and T2.
OHRQoL of participants storing their removable retainers in dry and wet conditions | 6 months
  The questionnaire is modified following a similar study of a randomised crossover clinical study comparing vacuum-formed thermoplastic retainers constructed on a conventional stone models and on 3D reconstructed study model.
  The OHRQoL is measured by using a modified 14-item Malaysian version of the Oral Health Impact Profile [OHIP-14(M)].
  The content focuses on the impact of oral health on quality of life through seven domains: 1) functional limitation, 2) physical pain, 3) psychological discomfort, 4) physical disability, 5) psychological disability, 6) social disability, and 7) handicap. Likert scale is used to measure the score for the responses; 0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, 4 = very often.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Postgraduate Clinic, Faculty of Dentistry, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn HW, Ha HR, Lim HN, Choi S. Effects of aging procedures on the molecular, biochemical, morphological, and mechanical properties of vacuum-formed retainers. J Mech Behav Biomed Mater. 2015 Nov;51:356-66. doi: 10.1016/j.jmbbm.2015.07.026. Epub 2015 Aug 3. PMID 26282078
- [Result] Ahn HW, Kim KA, Kim SH. A new type of clear orthodontic retainer incorporating multi-layer hybrid materials. Korean J Orthod. 2015 Sep;45(5):268-72. doi: 10.4041/kjod.2015.45.5.268. Epub 2015 Sep 23. PMID 26445722
- [Result] Al Groosh DH, Bozec L, Pratten J, Hunt NP. The influence of surface roughness and surface dynamics on the attachment of Methicillin-Resistant Staphylococcus aureus onto orthodontic retainer materials. Dent Mater J. 2015;34(5):585-94. doi: 10.4012/dmj.2014-045. PMID 26438981
- [Result] Alassiry AM. Orthodontic Retainers: A Contemporary Overview. J Contemp Dent Pract. 2019 Jul 1;20(7):857-862. PMID 31597809
- [Result] Chagas AS, Freitas KMS, Cancado RH, Valarelli FP, Canuto LFG, Oliveira RCG, Oliveira RCG. Level of satisfaction in the use of the wraparound Hawley and thermoplastic maxillary retainers. Angle Orthod. 2020 Jan;90(1):63-68. doi: 10.2319/031319-197.1. Epub 2019 Jul 22. PMID 31335161
- [Result] Fang J, Wang C, Li Y, Zhao Z, Mei L. Comparison of bacterial adhesion to dental materials of polyethylene terephthalate (PET) and polymethyl methacrylate (PMMA) using atomic force microscopy and scanning electron microscopy. Scanning. 2016 Nov;38(6):665-670. doi: 10.1002/sca.21314. Epub 2016 Mar 15. PMID 26991988
- [Result] Farhadian N, Usefi Mashoof R, Khanizadeh S, Ghaderi E, Farhadian M, Miresmaeili A. Streptococcus mutans counts in patients wearing removable retainers with silver nanoparticles vs those wearing conventional retainers: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2016 Feb;149(2):155-60. doi: 10.1016/j.ajodo.2015.07.031. PMID 26827971
- [Result] Kolenbrander PE, Andersen RN, Blehert DS, Egland PG, Foster JS, Palmer RJ Jr. Communication among oral bacteria. Microbiol Mol Biol Rev. 2002 Sep;66(3):486-505, table of contents. doi: 10.1128/MMBR.66.3.486-505.2002. PMID 12209001
- [Result] Littlewood SJ, Millett DT, Doubleday B, Bearn DR, Worthington HV. Retention procedures for stabilising tooth position after treatment with orthodontic braces. Cochrane Database Syst Rev. 2016 Jan 29;2016(1):CD002283. doi: 10.1002/14651858.CD002283.pub4. PMID 26824885
- [Result] Marsh PD. Dental plaque as a biofilm and a microbial community - implications for health and disease. BMC Oral Health. 2006 Jun 15;6 Suppl 1(Suppl 1):S14. doi: 10.1186/1472-6831-6-S1-S14. PMID 16934115
- [Result] Saub R, Locker D, Allison P, Disman M. Cross-cultural adaptation of the Oral Health Impact Profile (OHIP) for the Malaysian adult population. Community Dent Health. 2007 Sep;24(3):166-75. PMID 17958078